CLINICAL TRIAL: NCT05905380
Title: Analysis of the Efficacy and Tolerance of Covid-19 Convalescent Plasma and Monoclonal Antibodies in the Treatment of SARS-Cov2 Infections in Immunocompromised Patients
Brief Title: Covid-19 Convalescent Plasma and Monoclonal Antibodies Treatment of Immunocompromised Patients
Acronym: Covid-IC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8784
Record Dates: First submitted 2023-06-14; First posted 2023-06-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Convalescent Plasma Treatment
Keywords: Covid-19; SARS-Cov2; Immunosuppression; Cytokine; Convalescent Plasma; Monoclonal; Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on the use of convalescent plasma in the treatment of covid-19 are scarce: the results of randomized studies involving mainly immunocompetent patients are disappointing, while case series or retrospective data on more selected patients , in particular immunocompromised patients suggest a benefit in these patients whose clinical manifestation seems essentially related to the uncontrolled infection and not the cytokine storm.

ELIGIBILITY:
Inclusion criteria:

* Adult patient
* Immunocompromised patient (solid neoplasia, malignant hemopathy, solid organ transplantation, primary immune deficiency, systemic disease, chronic inflammatory disease, etc.)
* Hospitalized between 25/02/2020 and 15/01/2023 at HUS, ICANS, CH Colmar and CH Mulhouse
* Having received curative monoclonal antibody treatment or convalescent plasma treatment for SARS-Cov2 infection
* Patient who has not expressed, after being informed, his opposition to the reuse of his data for scientific research purposes.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient immunocompromised patient hospitalized between 25/02/2020 and 15/01/2023
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of the tolerance of Covid-19 convalescent plasma and monoclonal antibodies in the treatment of SARS-Cov2 infections in immunocompromised patients | Files analysed retrospectively from February 25, 2020 to January 15, 2023 will be examined
  This is a retrospective study on patient data from medical records from February 25, 2020 to January 15, 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France